CLINICAL TRIAL: NCT05218252
Title: Reliability and Versatility of Posterior Interosseous Artery Flap in Reconstructing Hand Soft Tissue Defects.
Brief Title: Reconstruction of Hand Soft Tissue Defects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed Talaat Ahmed, Principal investigator, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-01-06
Record Dates: First submitted 2022-01-17; First posted 2022-02-01 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Hand Injuries
Keywords: Posterior interosseous artery flap; Hand soft tissue defects
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hand soft tissue defects (Other): Patients with mild to moderate hand soft tissue defects with exposed bone, tendons or cartilage resulting from trauma, tumor ablation or postburn deformities.
  Interventions: Procedure: Posterior interosseous artery flap

INTERVENTIONS:
Procedure: Posterior interosseous artery flap — The use of distally based posterior interosseous artery flap from the forearm in reconstructing mild to moderate hand soft tissue defects

SUMMARY:
Evaluation of distally based posterior interosseous artery flap in reconstructing hand soft tissue defects that may result from trauma, extensive burns, tumor resection or congenital deformities.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with complex defects over the dorsal and palmar aspect of the wrist and the hand up to the proximal interphalangeal joint level, the whole thumb, and the first web space.
2. Small to moderate hand defects resulting from post-traumatic raw areas, post-traumatic deformities, postburn deformities and scar, post tumor resection, and congenital hand deformity.
3. Availability of a healthy donor site.

Exclusion Criteria:

1. Patients with a major uncontrollable medical illness.
2. Chronic heavy smokers.
3. Traumatic injury to the donor site.
4. Complex defects of the hand beyond the PIP joint level.

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2022-07 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Functional and aesthetic outcomes of posterior interosseous artery flap | 5 months from the end of treatment
  All patients will be evaluated with objective (functional) and subjective (aesthetic) criteria. Hand functionality will be evaluated using the disability of the arm, shoulder, and hand (DASH) score. The DASH score comprises 30 questions, and the score ranges from 30 points, for no limitation, to 150 points, for maximum limitation.
  The outcomes will be aesthetically reviewed with scar assessment measured as being good, fair, and poor. This assessment is subjective. Donor site problems are identiﬁed as cold intolerance, numbness, and pain. These will be evaluated as being either present in the patient or non-existent.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Talaat, Principal Investigator — Sohag University
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No